CLINICAL TRIAL: NCT01541384
Title: Medication Adherence in Kidney Transplant Recipients Using Automated Reminders and Provider Notification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 814788; K23DK078688 (NIH)
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Medication Adherence
Keywords: Kidney transplant; Adherence; Electronic pill bottles
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Medication Dosage Reminders (Experimental): Subject will receive electronic pill bottle that will track adherence. They will also be able to activate available dosage reminders (text message, phone message, email).
  Interventions: Device: Vitality GlowCaps
- Medicaiton Dosage Reminders + Coordinator Support (Experimental): Subject will receive electronic pill bottle that will track adherence. They will also be able to activate available dosage reminders (text message, phone message, email). The study coordinator will also check adherence every 2 weeks and alert the transplant team when it drops below 90%. The transplant team will determine the next best course of action.
  Interventions: Device: Vitality GlowCaps
- Usual Care with GlowCap (Other): Subject will receive electronic pill bottle that will track adherence but all reminders will be deactivated.
  Interventions: Device: Vitality GlowCaps

INTERVENTIONS:
Device: Vitality GlowCaps — The main research instrument is an electronic pill bottle called GlowCaps that has the ability to transmit reminder messages via email, text, and phone to the subject, and adherence data to special servers. The messages will be sent twice a day, if a subject misses a dose of their immunosuppression medication (tacrolimus). Each time the pill bottle is opened (or not opened), a date- and time-stamped wireless signal is sent to the Vitality server via the AT&T cellular network. No extra cellular or wireless service is required from subjects for the GlowCap to function.
  Note: GlowCaps are a "Class 1" Medical Device registered with the FDA. Because of this Class 1 designation, they are not subject to FDA testing or approval.

SUMMARY:
Novel wireless technology has created inexpensive tools that allow both accurate monitoring of adherence to pills as well as real-time interventions such as automated reminders in the event of a missed dose. In this study, the investigators will use Vitality GlowCaps, an electronic pill bottle. These pill bottles provide an unbiased assessment of pill bottle opening and a valid approach to verifying self-administered pill taking, reflecting not only daily use but also patterns of drug use and timing. At the prescribed times, bottle will electronically transmit whether a subject opened the pill cap to take the immunosuppressant medication via a built-in transmitter to the central server. The investigators will randomize participants to usual care, customized reminders, and customized reminders paired with provider notification in the event of low adherence.

The investigators' aim: To improve immunosuppression (IS) medication adherence in kidney transplant recipients.

The investigators' hypotheses: a) Automated reminders will improve adherence to immunosuppression compared to usual care, and b) Automated reminders, paired with provider notification about patients with poor adherence, will improve adherence to immunosuppression compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older) kidney or kidney-pancreas transplant recipient
* Hospital of the University of Pennsylvania (HUP) kidney transplant recipient (KTR)
* Recruitment within 2 weeks of discharge date
* Living within 120 miles of HUP

Exclusion Criteria:

* Vulnerable populations
* HIV seropositive status
* Poor English communication (which might hinder necessary communication with study coordinators)
* Discharge to care facility that handles patient medications
* Demonstrates inability or unwillingness to manage own medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter P Reese, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829

RESULTS

PARTICIPANT FLOW:
Groups:
- Medication Dosage Reminders: Subject will receive electronic pill bottle that will track adherence. They will also be able to activate available dosage reminders (text message, phone message, email).
  Electronic pill bottle: The main research instrument is an electronic pill bottle called GlowCaps that has the ability to transmit reminder messages via email, text, and phone to the subject, and adherence data to special servers. The messages will be sent twice a day, if a subject misses a dose of their immunosuppression medication (tacrolimus). Each time the pill bottle is opened (or not opened), a date- and time-stamped wireless signal is sent to the Vitality server via the AT&T cellular network. No extra cellular or wireless service is required from subjects for the GlowCap to function.
- Medicaiton Dosage Reminders + Coordinator Support: Subject will receive electronic pill bottle that will track adherence. They will also be able to activate available dosage reminders (text message, phone message, email). The study coordinator will also check adherence every 2 weeks and alert the transplant team when it drops below 90%. The transplant team will determine the next best course of action.
  Electronic pill bottle: The main research instrument is an electronic pill bottle called GlowCaps that has the ability to transmit reminder messages via email, text, and phone to the subject, and adherence data to special servers. The messages will be sent twice a day, if a subject misses a dose of their immunosuppression medication (tacrolimus). Each time the pill bottle is opened (or not opened), a date- and time-stamped wireless signal is sent to the Vitality server via the AT&T cellular network. No extra cellular or wireless service is required from subjects for the GlowCap to function.
- Usual Care With GlowCap: Subject will receive electronic pill bottle that will track adherence but all reminders will be deactivated.
  Electronic pill bottle: Device will remotely track adherence but reminders/alerts are deactivated.
Period: Overall Study
Arm/Group | Medication Dosage Reminders | Medicaiton Dosage Reminders + Coordinator Support | Usual Care With GlowCap
Started | 40 | 40 | 40
Completed | 40 | 39 | 38
Not Completed | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medication Dosage Reminders | Medicaiton Dosage Reminders + Coordinator Support | Usual Care With GlowCap | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12) | 50 (11) | 49 (11) | 50 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 16 | 48
  Male | 25 | 23 | 24 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 19 | 14 | 15 | 48
  White | 18 | 24 | 23 | 65
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 40 | 120

OUTCOME MEASURES:

1. Primary Outcome: Immunosuppression (Tacrolimus) Adherence
Description: The primary outcome will be the percentage of tacrolimus doses taken as directed during the final 90 days of this 180 day trial as measured by the GlowCap. This includes a 14 day "wash-in" period for device acclimatization.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: percentage of correct tacrolimus doses
Arm/Group | Medication Dosage Reminders | Medicaiton Dosage Reminders + Coordinator Support | Usual Care With GlowCap
Number analyzed (Participants) | 40 | 39 | 38
percentage of correct tacrolimus doses | 78 (14) | 88 (13) | 55 (17)

ADVERSE EVENTS:
Arm/Group | Medication Dosage Reminders | Medicaiton Dosage Reminders + Coordinator Support | Usual Care With GlowCap
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
The study did not assess clinical end points. Participants and study coordinators were not blinded to intervention arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No